CLINICAL TRIAL: NCT05985148
Title: A Phase I Dose Escalation Trial for Treatment of Chronic Thoracoabdominal Wall Pain Through Ablation of the Dorsal Spinal Nerve Using Single-Fraction Stereotactic Radiosurgery
Brief Title: A Study of Stereotactic Radiosurgery (SRS) to Treat Pain in the Chest and/or Stomach Wall
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-176
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Thoracoabdominal Wall Pain; Secondary to Parietal Pleura or Parietal Peritoneum Disease
Keywords: Stereotactic Radiosurgery (SRS); Ablation of the Dorsal Spinal Nerve; 22-176

STUDY DESIGN:
Intervention Model Description: This is a phase I clinical trial investigating the use of frameless single-fraction stereotactic radiosurgery (SRS) to treat chronic unilateral thoracoabdominal wall pain limited in distribution to three or fewer spinal levels from T3-T11 through ablation of the dorsal spinal nerve root.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-fraction stereotactic radiosurgery (SRS) (Experimental): Patients will be treated with single-fraction radiation therapy at three dose levels:
  70 Gy, 80 Gy, and 90 Gy using image-guided SRS techniques.
  Interventions: Radiation: Single-fraction stereotactic radiosurgery (SRS)

INTERVENTIONS:
Radiation: Single-fraction stereotactic radiosurgery (SRS) — Patients will be treated with single-fraction radiation therapy at three dose levels:
  70 Gy, 80 Gy, and 90 Gy using image-guided SRS techniques.

SUMMARY:
The researchers are doing this study to find out whether stereotactic radiosurgery (SRS) is a safe, practical (feasible), and effective treatment for people with chronic TAWP. The researchers will test different doses of SRS to find the highest dose that causes few or mild side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented history of chronic (≥ 3 months) thoracoabdominal wall pain (TAWP) attributable to ≤ 3 unilateral spinal levels as confirmed by diagnostic paravertebral nerve block or TENS (if results of the paravertebral nerve block are inconclusive) performed by an attending anesthesiologist specializing in pain management prior to study enrollment.
* Patients must have TAWP that is inadequately relieved by a trial of conventional pharmacologic therapy (defined as NRS pain score ≥ 4/10 while on treatment with conventional pharmacologic therapy for analgesia) as determined by an attending physician specializing in pain management.
* KPS ≥ 60%
* Age ≥ 18 years old

Exclusion Criteria:

* Patients with a life expectancy of < 6 months as predicted by the Adult Comorbidity Index (ACE-27, see Appendix 1)
* Patients with active autoimmune connective tissue disease
* Patients with bilateral TAWP
* Patients with preexisting pneumothorax
* Patients with preexisting excessive pleural effusion (extending > 3 vertebral levels)
* Systemic chemotherapy delivered or planned to be delivered within +/- 5 days of SRS
* Unable to undergo a diagnostic paravertebral nerve block
* Unable to undergo at least one of either a myelogram or spine MRI
* Patients for whom external beam treatment plans to deliver the prescription SRS dose to the lesion of interest cannot be safely designed as specified by the Dose Constraint Guidelines in Appendix 2

  * Evaluation of any radiation doses previously delivered to spinal cord/cauda equina and other critical structures (bowel, esophagus, lungs, kidneys, rectum) will be taken into consideration
  * If radiation dose from SRS would exceed any normal tissue constraint as noted in Appendix 2, the patient will be ineligible
* Abnormal complete blood count. Any of the following:

  * Platelet count < 75 K/µL
  * Hgb level < 9 g/dl
  * WBC < 3.5 K/µl
* Abnormal coagulation profile: INR > 2.5 INR and/or APTT > 80 seconds. Patients who are on anticoagulation medication that may not be safely held for the myelogram procedure (≥ 5 days for antiplatelet agents and warfarin; ≥ 24 hours for low-molecular weight heparin formulations) will be excluded.
* Allergy to local anesthestics
* Local infection at the site of injection of anesthetic
* Severe spinal deformities with anatomic distortion (severe scoliosis/kyphoscoliosis)
* Severe respiratory disease (i.e. oxygen dependent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
can be escalated from 70 Gy to 90 Gy without excessive DLTs | 2 years
  DLT's CTCAE grade ≥ 3 toxicity. Acute and late toxicity will be assessed by investigators and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Toxicities that cannot be graded using the Common Toxicity Criteria will be graded as 1 (mildly symptomatic), 2 (moderately symptomatic but not interfering significantly with function), 3 (causing significant interference with function), or 4 (life-threatening).

CONTACTS AND LOCATIONS:
Overall Officials: Josh Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm